CLINICAL TRIAL: NCT03926390
Title: Effect of Bovine Colostrum On T-Regulatory Cells, Prevention Of Late Onset Sepsis And Necrotizing Enterocolitis In Preterm Neonates
Brief Title: Gut Priming With Oral Bovine Colostrum for Preterm Neonates; Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ismail, Clinical professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU 50 / 2017
Record Dates: First submitted 2018-11-08; First posted 2019-04-24 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Late Onset Neonatal Sepsis; Necrotizing Enterocolitis of Newborn; Feeding; Difficult, Newborn
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non bovine colostrun (No Intervention): Preterm received preterm formula
- Bovine colostrum group (Active Comparator): Preterm received bovine colostrum as trophic feeding
  Interventions: Dietary Supplement: Bovine colostrum

INTERVENTIONS:
Dietary Supplement: Bovine colostrum — bovine colostrum for first 2 weeks
  Arms: Bovine colostrum group

SUMMARY:
The aim was to assess the ability of bovine colostrum concentrate to reduce the incidence of late-onset sepsis episodes and necrotizing enterocolitis in artificially fed preterm neonates and its effect on T regulatory cells. And to evaluate the effect of bovine colostrum concentrate on feeding tolerance, growth, hospital stay and mortality in preterm neonates.

DETAILED DESCRIPTION:
The study was interventional, double blinded and randomized trial ، performed on preterm neonates( <34 week) admitted on Ain ShamsUniversity (ASU) neonatal intensive care units (NICU) after considering exclusion criteria.

The enrolled patients was subdivided into two groups; group A are infants with non bovine colstrum and group B with bovine colostrum All infants received the standard neonatal care and underwent follow-up from birth until reach 37 week corrected gestational age, discharge or death whichever came first.

I. Data Collection: Careful history taking

1. Antenatal history including: rupture of membrane, Chorioamnionitis, history of urinary tract infection.
2. Natal history including: mode of delivery, place of delivery, the need for resuscitation, recorded Apgar score at 1minute and 5 minutes.
3. Postnatal history including: age of admission in neonatal intensive care unit, symptoms suggest infection.

II. Thorough clinical assessment:

1. Weight and Occiptofrontal circumference (twice weekly).
2. Complete examination including cardiovascular, respiratory, abdominal and neurological examination.

III. Laboratory investigations:

1. Complete blood picture, C-reactive protein on admission and repeated twice weekly
2. Blood culture before starting treatment and with any suspected sepsis.
3. In first 24 hours and the end of second week : Collecting peripheral blood mononuclear cells to be analyzed for cellular parameters by flow cytometry (CD4 T cells, CD25 L, FOXP3). Three subsets of CD4+ T cells will be defined according to CD25 staining: CD25- , CD25 low, and CD25 high. Cells expressing CD25 high will be chosen and gated for the detection of FOXP3+ T cells.

IV. Radiological investigations:

Chest X-ray (It was done on admission and repeated when needed). Abdominal X-ray (when necrotizing enterocolitis is suspected). Abdominal ultrasound (when necrotizing enterocolitis is suspected).

V. Follow-up and end-point of the study:

All infant underwent follow-up from birth until reach 37 week corrected gestational age, discharge or death whichever came first.NPO for more than 24 hours

The following primary outcome data was recorded:

* Clinical examination and laboratory investigations when clinically indicated for evidence of sepsis.
* Clinical examination and radiological investigations when clinically indicated for evidence of NEC.

A secondary outcome measure includes weight increment per kg per week, duration of hospitalization, mortality if any, monitoring adverse effects of treatment (if any); such as emesis, increased gastric residuals, increased abdominal girth, diarrhea, skin rash. Long term outcome includes necrotizing enterocolitis, and intracranial hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* • Preterm Neonate having a gestational age equal or less than 34 weeks at birth, admitted in Ain-Shams University NICUs

Exclusion Criteria:

* • Maternal risk factor of early onset sepsis, chorioamnionitis.

  * Proved early onset sepsis.
  * Life-threatening congenital abnormalities.
  * Inborn error of metabolism.
  * Chromosomal aberrations.
  * Neonates with underlying gastrointestinal problems (such as GIT anomalies) that prevent enteral feeding.
  * Perinatal asphyxia.

Ages: 24 Hours to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Late Onset Sepsis in the three groups | From time of randomization to discharge from nicu or death whichever comes first
  Incidence of Late Onset Sepsis in the studied group measured by rodwell and tollner sepsis scoring system
The incidence of Necrotizing Enterocolitis in the three groups | From time of randomization to discharge from nicu or death whichever comes first
  Incidence of Necrotizing Enterocolitis in the three groups diagnosed according to bell's staging
The change of Active T regulatory cells In the three groups | Change from base line at randomization and after intervention by 1 week
  Active T regulatory cells diagnosed by cell CD 4 expressing CD 25 high or simultaneously CD 25 plus FOXP3

SECONDARY OUTCOMES:
Feeding intolerance is defined as presence of at least 3 consecutive days of any of the following:emesis, gastric residuals, diarrhea, blood in stools or abnormally enlarged bowel loops | From time of randomization to discharge from nicu or death whichever comes first
  Feeding intolerance
Neonatal mortality | From time of randomization to discharge from nicu or death whichever comes first
  Number of deaths in the study group
Duration of hospital stay | From time of randomization to discharge from nicu or death whichever comes first
  Duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Awad, Principal Investigator — professor of pediatrics Ain Shams university
Locations (1):
- Medicin, Giza, Abasseya, Egypt

IPD SHARING:
Plan to Share IPD: No
research protocol